CLINICAL TRIAL: NCT06397599
Title: Denture Adhesive is a Patient Advantageous or Prosthetic Failure During Adaption Period: Randomized Control
Acronym: denture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sharaf Mohamed Yahia, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 6785/5; asharaf Email (Other: cairo university)
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Dental
Keywords: Denture adhesives, quality of life and OHIP-EDENT
MeSH Terms: interventions — Dental Cements; Dentures

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- denture adhesive (Active Comparator): use denture adhesive
  Interventions: Other: denture adhesive
- non adhesive (Active Comparator): conventional denture without denture adhesive
  Interventions: Other: denture adhesive

INTERVENTIONS:
Other: denture adhesive — use of adhesive for completely edentulous
  Other Names: use of adhesive for denture

SUMMARY:
Introduction: the complete denture wearers mainly complain of decrease of denture retention which affects on patient's quality of life Objective: to evaluate oral health-related quality of life (OHRQoL) of denture adhesive for completely edentulous denture wearers.

Material and methods : 32 patients(new denture wearers) were selected form prosthdontic clinic in three dental faculties in various region in Egypt, there were 22 females (68%) and 10 males (46%) were distributed in two groups: conventional group without adhesive and adhesive group with adhesive application n = 16;, in a cross over study. evaluation by Oral Health Impact Profile in Edentulous Adults (OHIP-EDENT) inventory at 1, 2 and 3 months after the insertion of new complete dentures. Data were analyzed using 2-way ANOVA test and Generalized Estimating Equations (GEEs), α = 0.05.

DETAILED DESCRIPTION:
32 patients(new denture wearers) were selected form prosthdontic clinic in three dental faculties in various region in Egypt, there were 22 females (68%) and 10 males (46%) were distributed in two groups: conventional group without adhesive and adhesive group with adhesive application n = 16;, in a cross over study. evaluation by Oral Health Impact Profile in Edentulous Adults (OHIP-EDENT) inventory at 1, 2 and 3 months after the insertion of new complete dentures. Data were analyzed using 2-way ANOVA test and Generalized Estimating Equations (GEEs), α = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* completely edentulous

Exclusion Criteria:

* no

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
patients satisfaction | 6 months
  questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided